CLINICAL TRIAL: NCT06916598
Title: Consensus Statements on Definition, Components and Grading of Postoperative Pulmonary Complications- an International Delphi Study
Brief Title: Consensus Statements on Definition, Components and Grading of Postoperative Pulmonary Complications
Acronym: PrECiSIOn
Status: Enrolling by invitation | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: University of Wolverhampton (Other); The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Responsible Party: Principal Investigator, Prof. Dr. Marcus J. Schultz, Professor dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: PrECiSIOn
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-04

CONDITIONS: Postoperative Pulmonary Complications
Keywords: postoperative pulmonary complications; postoperative complications; postoperative pulmonary atelectasis; postoperative pulmonary care; outcomes assessment; Delphi study
MeSH Terms: conditions — Postoperative Complications; Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Delphi Panellists: An international panel of 35-40 panellists from Anesthesiology, Surgery or Intensive Care Medicine and including patient representatives, will be invited to this Delphi study. A concerted effort will be made to include panellists from low- and middle-income countries and both sexes.
  Interventions: Other: Delphi study
- Patient and Public involvement: Individuals who have either personally experienced PPCs following surgery within the last 5 years or, primary caregivers of such patients will be recruited as patient care representatives.
  Interventions: Other: Structured Interview

INTERVENTIONS:
Other: Delphi study — This Delphi study involves multiple iterative rounds until a stable consensus or dissensus is reached on all the statements.
  Groups: Delphi Panellists
Other: Structured Interview — Structured interviews will be conducted by members of the steering committee and an independent qualitative research expert. A pilot-tested case vignette along with a Likert scale-based questionnaire, will be employed to gather insights regarding the impact and severity of PPCs. The impact of the individual components of PPCs will be evaluated on a 7-point Global Rate of Change (GRC) scale (from "very much worse" to very much better") to calculate the minimal clinical important difference. Patient care representatives will be engaged in anonymous voting on the questionnaire. PPCs' rankings and key themes synthesised from the interviews will be shared with the panel in the second Delphi round, facilitating the integration of patient perspectives into the consensus process.
  Groups: Patient and Public involvement

SUMMARY:
An international team of experts is working on a project called PrECiSIOn to develop a clear, consistent definition of PPCs. The goals of this study are to:

* Define postoperative pulmonary complications in a way that makes sense for patients, families, and healthcare providers.
* Rank complications by severity so doctors can focus on the most serious ones first.
* Decide how and when to monitor patients after surgery to catch problems early.

DETAILED DESCRIPTION:
Postoperative pulmonary complications (PPCs) are associated with prolonged hospital stays, increased mortality, and significant clinical and economic burdens. Despite their importance, the definition of PPCs varies across studies, leading to inconsistencies in reported incidence rates and research outcomes. Existing definitions, such as the EPCO criteria, have been developed based on expert opinion but lack systematic consensus-building methods.

To address these limitations, the StEP collaboration conducted a systematic review and Delphi process to refine PPC classifications. However, challenges remain, including the lack of universal definitions, hierarchical ranking of complications, and representation from diverse healthcare settings. Composite outcome measures improve statistical power but may obscure differences in severity and clinical significance among PPC subtypes.

The PrECiSIOn Delphi initiative aims to develop an expert consensus on defining PPCs, grading their severity, and determining standardized monitoring methods. The goal is to create a valid, reliable, and universally accepted patient-centered definition of PPCs that enhances comparability across studies and informs clinical decision-making.

ELIGIBILITY:
Inclusion Criteria: Panellists will be identified based on either of the following criteria

* At least 10 years of clinical experience as a staff member in Anesthesiology, Surgery or Intensive Care Medicine with involvement in care of patients with postoperative complications
* Author of at least three publications (observational studies or randomised controlled trials) using postoperative pulmonary complications as a primary or secondary outcome For patients and public involvement Individuals who have either personally experienced PPCs following surgery within the last 5 years or, primary caregivers of such patients will be recruited as patient care representatives. Proficiency in English is required. To mitigate potential bias, patient care representatives mustn't maintain a professional or advisory relationship with the steering committee or panellists.

Exclusion Criteria

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: To encourage the continued engagement of the panellists and help prevent them from dropping out before completing the full process, at least three personalised email reminders will be sent during each Delphi round, in addition to an effort to establish personal contact. Furthermore, all panellists will be recognised as collaborative authors in the final publication in appreciation of their professional expertise. Should the attrition rate of panellists exceed 20%, a sensitivity analysis will be conducted, considering the plausible worst-case and best-case scenarios, and taking into account the opinions of non-responders.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Generate consensus on the postoperative pulmonary complications construct | 3-6 months
  A diverse group of panellists worldwide, based on pre-specified qualification criteria, will conduct iterative Delphi rounds to generate consensus on the construct of postoperative pulmonary complications.

SECONDARY OUTCOMES:
Generate consensus on the postoperative pulmonary complications definition and components | 3-6 months
  A diverse group of panellists worldwide, based on pre-specified qualification criteria, will conduct iterative Delphi rounds to generate consensus on the definition and components of postoperative pulmonary complications
Generate consensus on the on the timeframe of monitoring for postoperative pulmonary complications | 3-6 months
  A diverse group of panellists worldwide, based on pre-specified qualification criteria, will conduct iterative Delphi rounds to generate consensus on the timeframe of monitoring for postoperative pulmonary complications
Generate consensus on the methods of monitoring of postoperative pulmonary complications | 3-6 months
  A diverse group of panellists worldwide, based on pre-specified qualification criteria, will conduct iterative Delphi rounds to generate consensus on the methods of monitoring of postoperative pulmonary complications.
Generate consensus on weightage grade of individual postoperative pulmonary complications | 3-6 months
  A diverse group of panellists worldwide, based on pre-specified qualification criteria, will conduct iterative Delphi rounds to generate consensus on weightage grade of individual postoperative pulmonary complications.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Schultz, PhD, Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- New Cross Hospital, Wolverhampton, Wolverhampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The IPD is available to investigators and can be shared with appropriate requests.

REFERENCES:
- [Background] Myles PS, Grocott MP, Boney O, Moonesinghe SR; COMPAC-StEP Group. Standardizing end points in perioperative trials: towards a core and extended outcome set. Br J Anaesth. 2016 May;116(5):586-9. doi: 10.1093/bja/aew066. No abstract available. PMID 27106961
- [Background] Gottlieb M, Caretta-Weyer H, Chan TM, Humphrey-Murto S. Educator's blueprint: A primer on consensus methods in medical education research. AEM Educ Train. 2023 Jul 11;7(4):e10891. doi: 10.1002/aet2.10891. eCollection 2023 Aug. PMID 37448627
- [Background] Abbott TEF, Fowler AJ, Pelosi P, Gama de Abreu M, Moller AM, Canet J, Creagh-Brown B, Mythen M, Gin T, Lalu MM, Futier E, Grocott MP, Schultz MJ, Pearse RM; StEP-COMPAC Group. A systematic review and consensus definitions for standardised end-points in perioperative medicine: pulmonary complications. Br J Anaesth. 2018 May;120(5):1066-1079. doi: 10.1016/j.bja.2018.02.007. Epub 2018 Mar 27. PMID 29661384
- [Background] Jammer I, Wickboldt N, Sander M, Smith A, Schultz MJ, Pelosi P, Leva B, Rhodes A, Hoeft A, Walder B, Chew MS, Pearse RM; European Society of Anaesthesiology (ESA) and the European Society of Intensive Care Medicine (ESICM); European Society of Anaesthesiology; European Society of Intensive Care Medicine. Standards for definitions and use of outcome measures for clinical effectiveness research in perioperative medicine: European Perioperative Clinical Outcome (EPCO) definitions: a statement from the ESA-ESICM joint taskforce on perioperative outcome measures. Eur J Anaesthesiol. 2015 Feb;32(2):88-105. doi: 10.1097/EJA.0000000000000118. PMID 25058504
- [Background] Lusquinhos J, Tavares M, Abelha F. Postoperative Pulmonary Complications and Perioperative Strategies: A Systematic Review. Cureus. 2023 May 9;15(5):e38786. doi: 10.7759/cureus.38786. eCollection 2023 May. PMID 37303413
- [Background] Shander A, Fleisher LA, Barie PS, Bigatello LM, Sladen RN, Watson CB. Clinical and economic burden of postoperative pulmonary complications: patient safety summit on definition, risk-reducing interventions, and preventive strategies. Crit Care Med. 2011 Sep;39(9):2163-72. doi: 10.1097/CCM.0b013e31821f0522. PMID 21572323
- [Background] Canet J, Sabate S, Mazo V, Gallart L, de Abreu MG, Belda J, Langeron O, Hoeft A, Pelosi P; PERISCOPE group. Development and validation of a score to predict postoperative respiratory failure in a multicentre European cohort: A prospective, observational study. Eur J Anaesthesiol. 2015 Jul;32(7):458-70. doi: 10.1097/EJA.0000000000000223. PMID 26020123
- [Background] Piccioni F, Langiano N, Bignami E, Guarnieri M, Proto P, D'Andrea R, Mazzoli CA, Riccardi I, Bacuzzi A, Guzzetti L, Rossi I, Scolletta S, Comi D, Benigni A, Pierconti F, Coccia C, Biscari M, Murzilli A, Umari M, Peratoner C, Serra E, Baldinelli F, Accardo R, Diana F, Fasciolo A, Amodio R, Ball L, Greco M, Pelosi P, Della Rocca G; One-Lung Ventilation Investigators Group (Supplementary Appendix S1). One-Lung Ventilation and Postoperative Pulmonary Complications After Major Lung Resection Surgery. A Multicenter Randomized Controlled Trial. J Cardiothorac Vasc Anesth. 2023 Dec;37(12):2561-2571. doi: 10.1053/j.jvca.2023.04.029. Epub 2023 Apr 27. PMID 37730455
- [Background] Fernandez-Bustamante A, Frendl G, Sprung J, Kor DJ, Subramaniam B, Martinez Ruiz R, Lee JW, Henderson WG, Moss A, Mehdiratta N, Colwell MM, Bartels K, Kolodzie K, Giquel J, Vidal Melo MF. Postoperative Pulmonary Complications, Early Mortality, and Hospital Stay Following Noncardiothoracic Surgery: A Multicenter Study by the Perioperative Research Network Investigators. JAMA Surg. 2017 Feb 1;152(2):157-166. doi: 10.1001/jamasurg.2016.4065. PMID 27829093
- [Derived] Nasa P, Yurttas T, Battaglini D, Blot S, Fernandez-Bustamante A, Gama de Abreu M, van Meenen DM, Myatra SN, Serpa Neto A, Oppong R, Paulus F, Renukappa S, Schultz MJ, Slutsky AS, Hemmes SNT; PrECiSIOn-group. Consensus on the definition, components, timeframe and grading of composite outcome of postoperative pulmonary complication-protocol for an international mixed-method consensus study (PrECiSIOn). BMJ Open. 2025 Aug 19;15(8):e103888. doi: 10.1136/bmjopen-2025-103888. PMID 40829816